CLINICAL TRIAL: NCT00292708
Title: Randomized Multicenter Trial of Antibiotic Prophylaxis in Elective Colorectal Surgery: Single-Dose Vs. Three Doses of Second-Generation Cephalosporin
Brief Title: Trial of Antibiotic Prophylaxis in Elective Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C000000069
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2006-02-16 (Estimated); Status verified 2006-02

CONDITIONS: Colorectal Surgery
Keywords: Antibiotics; Prophylaxis; Surgical wound infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefmetazole; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Cefmetazole (drug)

SUMMARY:
To determine the optimal prophylactic antibiotics administration method in elective colorectal surgery

DETAILED DESCRIPTION:
Use of prophylactic antibiotics in elective colorectal surgery is essential. Although single-dose prophylactic antibiotics are recommended, the efficacy of single-dose cephalosporin without metronidazole and oral antibiotics is not fully proven. We conducted a multicenter randomized trial of single-dose vs. three doses of the second-generation cephalosporin, cefmetazole.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal diseases (cancer, large polyp, carcinoid, lymphoma,sarcoma and so on)
* Elective colorectal resection

Exclusion Criteria:

* Emergent operation
* Ileus
* No resection
* Preoperative infectious diseases
* Penicillin or cephalosporin allergy
* Antibiotics administration before surgery
* Inflammatory bowel diseases
* Angina or myocardial infarction
* Renal dysfunction
* Diabetes mellitus
* Steroid administration before surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-05; Study Completion 2005-07

PRIMARY OUTCOMES:
Incidence of incisional surgical site infection (SSI)

SECONDARY OUTCOMES:
Incidences of organ/space SSI and other infectious diseases. Other postoperative complications and postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Shin Fujita, MD. PhD., Principal Investigator — Japan National Cancer Center Hospital
Locations (7):
- Japan (7):
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - National Cancer Center East Hospital, Kashiwa
  - Nagoya Medical Center, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - National Cancer Center Hospital, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata

REFERENCES:
- [Derived] Fujita S, Saito N, Yamada T, Takii Y, Kondo K, Ohue M, Ikeda E, Moriya Y. Randomized, multicenter trial of antibiotic prophylaxis in elective colorectal surgery: single dose vs 3 doses of a second-generation cephalosporin without metronidazole and oral antibiotics. Arch Surg. 2007 Jul;142(7):657-61. doi: 10.1001/archsurg.142.7.657. PMID 17638804
- See also: UMIN Clinical Trial Registry: Unique trial number C000000069 — http://www.umin.ac.jp/ctr/index.htm